CLINICAL TRIAL: NCT04810793
Title: The Study on the Selection of Time for Retreatment of Helicobacter Pylori After Eradication Failure
Status: Completed | Type: Observational
Sponsor: Shandong University (Other)
Collaborators: Taian City Central Hospital (Other); Dezhou People's Hospital (Other); Weifang Medical University (Other); The Affiliated Hospital of Qingdao University (Other); Shengli Oilfield Hospital (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, Professor, Director of gastroenterology department of Qilu hospital, Shandong University
Other Study IDs: 2020-SDU-QILU-G101
Record Dates: First submitted 2021-03-21; First posted 2021-03-23 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Helicobacter Pylori
Keywords: Re-eradication time; Remedial treatment
MeSH Terms: interventions — Amoxicillin; Levofloxacin; Esomeprazole; Furazolidone; Tetracycline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Amoxicillin-Levofloxacin-Esomeprazole-containing quadruple group: Patients in amoxicillin-levofloxacin-esomeprazole-containing quadruple group will receive esomeprazole (Nexium) 40mg po bid, amoxicillin 1000mg po bid, bismuth potassium citrate(Lizhudele) 220mg po bid, and levofloxacin 500mg po qd for 14d.
  Interventions: Drug: Amoxicillin , Levofloxacin and Esomeprazole
- Amoxicillin-Furazolidone-Esomeprazole-containing quadruple group: Patients in amoxicillin-furazolidone-esomeprazole-containing quadruple group will receive esomeprazole (Nexium) 40mg po bid, amoxicillin 1000mg po bid, bismuth potassium citrate(Lizhudele) 220mg po bid, and furazolidone (Liteling) 100mg po bid for 14d.
  Interventions: Drug: Amoxicillin , Furazolidone and Esomeprazole
- Tetracycline-Furazolidone-Esomeprazole-containing quadruple group: Patients in tetracycline-furazolidone-esomeprazole-containing quadruple group will receive esomeprazole (Nexium) 40mg po bid, tetracycline 500mg po qid, bismuth potassium citrate(Lizhudele) 220mg po bid, and furazolidone (Liteling) 100mg po bid for 14d.
  Interventions: Drug: Tetracycline , Furazolidone and Esomeprazole
- Amoxicillin-Levofloxacin-Vonoprazan fumarate-containing quadruple group: Patients in amoxicillin-levofloxacin-vonoprazan fumarate-containing quadruple group will receive vonoprazan fumarate 20mg po bid, amoxicillin 1000mg po bid, bismuth potassium citrate(Lizhudele) 220mg po bid, and levofloxacin 500mg po qd for 14d.
  Interventions: Drug: Amoxicillin,Levofloxacin and Vonoprazan fumarate
- Amoxicillin-Furazolidone-Vonoprazan fumarate-containing quadruple group: Patients in amoxicillin-furazolidone-vonoprazan fumarate-containing quadruple group will receive vonoprazan fumarate 20mg po bid, amoxicillin 1000mg po bid, bismuth potassium citrate(Lizhudele) 220mg po bid, and furazolidone (Liteling) 100mg po bid for 14d.
  Interventions: Drug: Amoxicillin,Furazolidone and Vonoprazan fumarate
- Tetracycline-Furazolidone-Vonoprazan fumarate-containing quadruple group: Patients in tetracycline-furazolidone-vonoprazan fumarate-containing quadruple group will receive vonoprazan fumarate 20mg po bid, tetracycline 500mg po qid, bismuth potassium citrate(Lizhudele) 220mg po bid, and furazolidone (Liteling) 100mg po bid for 14d.
  Interventions: Drug: Tetracycline,Furazolidone and Vonoprazan fumarate

INTERVENTIONS:
Drug: Amoxicillin , Levofloxacin and Esomeprazole — Esomeprazole-Bismuth-Amoxicillin-Levofloxacin-containing quadruple regimens
  Groups: Amoxicillin-Levofloxacin-Esomeprazole-containing quadruple group
Drug: Amoxicillin , Furazolidone and Esomeprazole — Esomeprazole-Bismuth-Amoxicillin-Furazolidone-containing quadruple regimens
  Groups: Amoxicillin-Furazolidone-Esomeprazole-containing quadruple group
Drug: Tetracycline , Furazolidone and Esomeprazole — Esomeprazole-Bismuth-Tetracycline-Furazolidone-containing quadruple regimens
  Groups: Tetracycline-Furazolidone-Esomeprazole-containing quadruple group
Drug: Amoxicillin,Levofloxacin and Vonoprazan fumarate — Amoxicillin-Levofloxacin-Vonoprazan fumarate-containing quadruple group
  Groups: Amoxicillin-Levofloxacin-Vonoprazan fumarate-containing quadruple group
Drug: Amoxicillin,Furazolidone and Vonoprazan fumarate — Amoxicillin-Furazolidone-Vonoprazan fumarate-containing quadruple group
  Groups: Amoxicillin-Furazolidone-Vonoprazan fumarate-containing quadruple group
Drug: Tetracycline,Furazolidone and Vonoprazan fumarate — Tetracycline-Furazolidone-Vonoprazan fumarate-containing quadruple group
  Groups: Tetracycline-Furazolidone-Vonoprazan fumarate-containing quadruple group

SUMMARY:
The patients who accepted the quadruple eradication program of the helicobacter pylori but failed to eradicate helicobacter pylori will be assessed the most suitable re-eradication time of helicobacter pylori.

DETAILED DESCRIPTION:
Helicobacter pylori (HP) infection is a common global infectious disease, which is an important cause of chronic gastritis, peptic ulcer and gastric cancer.

At present, due to the non-standard Helicobacter pylori eradication program in clinical work, poor patient compliance and other reasons, the phenomenon of HP eradication treatment failure is more and more common. However, there is still no conclusion on the most appropriate time for remedial treatment in patients with Hp eradication failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients, aged between 18 and 70 years old, with positive H. pylori infection that was eradicated by previous therapies but failed are included. The H. pylori infection is confirmed by the positive rapid urease test or 13C-breath test.

Exclusion Criteria:

* Patients with significant underlying disease including liver, cardiac, pulmonary, and renal diseases, neoplasia, coagulopathy and genetic diseases, history of gastric surgery, pregnancy, breast-feeding, active gastrointestinal bleeding, the use of PPI, NSAID or antibiotics during the 4 weeks prior to enrolment, and previous history of allergic reactions to any of the medications used in this protocol. Patients previously treated with H. pylori eradication regimens or those unwilling to participate in the study were also excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients in Shandong province,aged between 18 and 70 years old, with positive H. pylori infection that was eradicated by previous therapies but failed are included.
Sampling Method: Probability Sample
Enrollment: 820 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
The most suitable re-eradication time | 1year
  The most suitable re-eradication time will be assessed by paired comparison method .

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, MD,PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China